CLINICAL TRIAL: NCT03995134
Title: Target Controlled Infusion Using Propofol and Remifentanil for Moderate Sedation in Dentistry
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00083505
Record Dates: First submitted 2019-06-17; First posted 2019-06-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2020-01

CONDITIONS: Sedative Adverse Reaction
Keywords: Use of propofol and remifentanil administered with TCI pump
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Propofol and Remifentanil: Procedural sedation in Dentistry provided by a Target Controlled Infusion pump using propofol as the sedative/hypnotic agent and Remifentanil as the opioid analgesic agent.
  Interventions: Combination Product: Propofol and Remifentanil administered by TCI pump

INTERVENTIONS:
Combination Product: Propofol and Remifentanil administered by TCI pump — Propofol, Remifentanil, Alaris PK (pharmacokinetic) infusion pump with TCI

SUMMARY:
The purpose of this university study is to evaluate the use of an advanced dental sedation technique involving two syringe-type pumps called Target Controlled Infusion (TCI) pumps. Two oral surgeons and a general dentist from New Zealand are assisting a Canadian research team as they study this intravenous sedation technique and its use in dental offices. This sedation technique is broadly used in other parts of the world and is known to reduce anxiety and discomfort during dental or medical procedures.

The New Zealand Dental Council and Health Canada have approved the drugs involved and the TCI pumps. In this study, one pump will be used to administer a sedative drug called propofol and the other to administer a pain-relief analgesic drug called remifentanil. The pumps and drugs are licensed in New Zealand and Canada and are not experimental.

These pumps are operated by special software modules that are specific to each drug, and a computer within the pump controls the pump operation allowing a stable and constant level of drug in the blood stream.

Your oral surgeon or dentist will titrate or add small amounts of drug till the you are quite relaxed before proceeding with your dental treatment. The dentist has overall control of the pump and the amount of drug given and can change the amount if it is too little or too much for you, or completely stop the pump if necessary for safety..

The TCI sedation, including your dental treatment will be conducted by two oral surgeons and a general dentist in their respective New Zealand dental offices. Each clinician is well trained and experienced with this form of sedation.

DETAILED DESCRIPTION:
Purpose:

Moderate (conscious) sedation is a common pharmacological approach to managing psychological anxiety and physical pain associated with dental procedures including surgery. While maintaining patient responsiveness to verbal and tactile stimuli, safety of conducting moderate sedation in dental clinic is well documented with infrequent complications. Preferred drug choices for administering moderate intravenous (i.v.) sedation are midazolam (benzodiazepine sedative) and fentanyl (opioid analgesic) because their safety and efficacy have been well established and are currently considered the Standard of Care (SoC) worldwide.

The use of drugs intended for general anesthesia to provide moderate (conscious) sedation is increasingly being considered for dental sedation as there are a number of benefits when compared to the SoC. For example, propofol has a favorable pharmacokinetic profile and absence of lingering side-effects; drugs (propofol and remifentanil) with fast onset and offset times are most useful for balancing adequate hypnosis/analgesia with rapid recovery.

This clinical research study will explore the potential benefits of controlled administration of propofol (hypnotic agent) and remifentanil (opioid analgesic agent) utilizing two Target Controlled Infusion (TCI) pumps for moderate i.v. sedation by a sedationist/operator in a dental office-based environment.

Standardized care for moderate (conscious) sedation is guided by the following principle:

Drugs and techniques used to provide moderate (conscious) sedation for dental treatment should carry a margin of safety wide enough to render loss of consciousness unlikely.

The level of sedation must be such that the patient remains conscious and is able to both understand and respond to verbal commands either alone or accompanied by light tactile stimulus; Modified Ramsay Sedation score of 3 or 4 .

The current SoC for i.v. dental sedation in Canada and New Zealand is the administration of a single benzodiazepine agent alone or in combination with an opioid analgesic agent to achieve moderate or conscious sedation whereby the patient responds to voice or light tough stimulus throughout the procedure.

The purpose of this study is to explore the advantages/disadvantages and risks/benefits of TCI interventional sedation technique in an dental office-based environment.

Hypothesis:

Increasingly, the controlled use of propofol and remifentanil utilizing pharmacokinetic programmed syringe pumps called Target Controlled Infusion (TCI) pump are being considered as an alternative option for dental sedation for the operator/sedationist and their sedation team. Is this sedation technique a viable option to the SoC?

Within the TCI system, specific pharmacokinetic algorithms have been developed for each drug, accounting for drug distribution, elimination, and metabolism, thus providing a stable, constant concentration of drug at the plasma (blood) or brain level. The drugs used are short acting, thus the clinician can quickly titrate the drugs to the desired sedative effect and if necessary can incrementally increase or decrease the drug's sedative/analgesic effect to meet patient's needs and procedural stimulus. In sum, the short-acting nature of the drugs, combined with a specified delivery algorithm have the potential in allowing better patient care in dental office setting through adapting dosage to patient needs, thus allowing better control, a shorter recovery time with early home readiness.

Justification:

Adequacy of procedural sedation depends on the maintenance of brain propofol and remifentanil concentrations which are clinically appropriate and in equilibrium with levels in the plasma. The best way to achieve this state is from TCI dedicated pharmacokinetic pumps. These devices solve the complex equations which describe the distribution of agents between compartments and allow for rapid adjustments in targets to achieve the desired clinical effect.

Health Canada has approved the use of propofol and remifentanil for on-label use for dental sedation and anesthesia, and has approved the Alaris PK infusion pump with TCI for use in Canada. New Zealand Dental Council has also approved and permitted propofol and remifentanil and the Alaris PK infusion pump for dental sedation.

American Society of Anesthesiologist's Moderate Sedation Guidelines 2018 provides guidance and recommendations that include sedative/analgesic medications intended for general anesthesia (propofol and remifentanil) can also be safely administered for moderate sedation across health professions and environments.

A published research study exploring the use of TCI pump technology in medicine to the year 2015, conservatively estimated the following:

* Use worldwide >90 countries.
* TCI pump sales >60,000 units.
* Anesthesia and sedation >20 million administrations.
* Commercial usage of TCI process >2 decades in clinical use.

Dr. Lobb is unaware of:

* Any dentist/dental specialist in Canada using propofol and remifentanil with TCI technology for moderate sedation.
* Any dental college in Canada that has issued a permit to use propofol and remifentanil with TCI technology for moderate sedation.
* Any Canadian university involved in clinical research using propofol and remifentanil with TCI technology for dental sedation.

Thus, to advance important and relevant Canadian clinical research in the administration of propofol and remifentanil with TCI pumps for sedation dentistry, Dr. Lobb has invited dental experts outside of Canada to partner with a research team from the University of Alberta. The following reasons justifies this rationale:

Oral surgeons in New Zealand have been world leaders in the use of TCI sedation in dentistry for over a decade. The two pump TCI sedation process has become a Standard of Care in a number of dentist/dental specialist offices.

The New Zealand dental group licensed to administer propofol and remifentanil with TCI pump technology includes oral surgeons, oral and maxillofacial surgeons and general dentists, with:

* >10 years' experience with TCI sedation.
* >40,000 collective administrations.
* Two New Zealand oral surgeons and a general dentist have consented to participate in this clinical research study. All three are experienced TCI sedation practitioners.
* The clinical phase of this research study will be completed within their respective dental practice facilities in New Zealand.
* he population numbers and demographic profile of New Zealand is quite similar to Alberta.
* The type of dental surgery and general dentistry performed in New Zealand is similar in scope to that practiced by Alberta dental practitioners.

Objectives:

The overall objective of the research is to validate a sedation technique that is proposed to be more controllable and less intrusive to patients. Specifically, in this prospective pilot study, we seek to determine the safety, effectiveness, and comparability of the controlled administration of propofol and remifentanil utilizing two TCI syringe pumps for moderate sedation in dentistry through establishing, identifying, and refining a study protocol in this pilot study in preparation for a larger study, or a replication study in Canada.

Research Methods/Procedures:

This is a prospective, pilot study, with the TCI sedation and clinical component of the study being completed by two oral surgeons and one general dentist in New Zealand. The rationale for having the sedation and clinical treatment performed in New Zealand is there are no dentists/dental specialists licensed by the Alberta Dental Association and College to use this form of i.v. sedation in Alberta at this time.

All treatment will occur at the oral surgery offices of Drs. Don Macalister and David Chrisp in Auckland and Taruanga respectively, and general dental office of Dr. Graham Shaw in Auckland, New Zealand.

A total of 100 patients are the requirement for this pilot study across three sites. This study will be of nine months' duration, from September 1, 2018 to June 30, 2019, or when 40 patients have been successfully recruited to the study at each site oral surgery site and 20 at the general dentistry site.

Intravenous sedation study participants will receive the established TCI dental i.v. sedation consistent to each oral surgeon and general dentist office protocol.

The participating oral surgeons/dentist will abide by any research protocols established by the New Zealand Ethics Office, and the University of Alberta, Research Ethics Office.

During the sedation: the use of appropriate physiologic and electronic monitoring, standardized intravenous administration sets, TCI infusion pumps, personnel, record keeping and discharge criteria will be used. Brain function monitoring (pEEG) provides additional information to the clinician during titration of propofol and remifentanil.

Post-sedation, all patients are followed up with a phone call and if there are any concerns, the patients will be seen immediately. In the event of any problems or concerns after hours, the phone number of the oral surgeon/dentist is available on the post-sedation instruction sheet.

Immediately following the sedation and prior to discharge, the participants will be asked a series of questions from the patient satisfaction questionnaire. In the follow-up portion of the study, participants will be asked the same series of questions from the patient satisfaction questionnaire; 24 - 48 hours following the sedation.

TCI sedation involves the use of controlled administration of propofol and remifentanil utilizing two TCI pumps (Alaris PK infusion pump with TCI). The software models used in New Zealand differ slightly from that currently available in Canada. In New Zealand effect-site or brain level software (Schnider for propofol and Minto for remifentanil) will be used.

In Canada, the licensed software for the same pump is plasma level software (Marsh for propofol and Minto for remifentanil).

The propofol TCI models (Schnider or Marsh) prove highly effective in combination with remifentanil TCI. Clinical practice demonstrates there is no 'best' TCI model for propofol. The clinician should become familiar with the model which matches the patient characteristics of their usual patient population. Regardless of pharmacokinetic model used, clinical monitoring of the patient remains an important and integral part of the sedation team's role and patient care.

The dental procedures will be what is normally performed in each New Zealand office, and the scope of these procedures is similar to that performed by dental practitioners in Alberta.

Plan for Data Analysis:

Independent t-test and analysis of covariance will be used to compare differences in safety and effectiveness measures as described. Box M test will be used to evaluate comparability of variance between sites. A statistical covariate will also be used to conduct comparison of results taking account of the risk associated with patient demographics.

Data collected from patients will first be processed such that values across multiple time-points, collected through survey and patient record, will reflect as one record.

Incomplete or problematic records will be removed from the analysis. Descriptive statistics will be presented for all measures of secondary objectives, confidence interval estimates, proportion and statistical tests will be conducted to evaluate safety and effectiveness findings.

ELIGIBILITY:
Inclusion Criteria:

* Patient age: ≥18 years of age.
* Patients who are generally healthy (American Society of Anesthesiology [ASA] Physical Status I), or patients with mild systemic disease (ASA Patient Physical Status II).
* Both genders eligible.

Exclusion Criteria:

* Patients who would normally be unsuitable candidates for treatment in non-hospital dental facilities undergoing intravenous sedation.
* Medically complex or unwell patients who may require medical anesthesiologist or hospital assistance, i.e., ASA III or greater.
* Patients with a history of anesthetic-related complications or difficult airway management that may require the assistance of an anesthesiologist.
* Patients allergic to propofol or fentanyl compounds.
* Patients who are unable to, or refuse to sign the consent form.
* Female patients who are pregnant, or suspect they may be.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: New Zealand citizens
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2019-08-03 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
Maintaining Patient Responsiveness during Target Controlled Infusion sedation | 5 minute
  Number of participants with treatment-related adverse events as assessed by loss of consciousness or responsiveness

SECONDARY OUTCOMES:
Rates of adverse events and side effects when using TCI for Procedural Sedation in Dentistry - oxygen desaturation | Baseline and 5 minute
  Sum of time intervals of oxygen desaturation below SpO2 of 90.
Rates of adverse events and side effects when using TCI for Procedural Sedation in Dentistry - blood pressure | Baseline and 5 minute
  A change of Mean Arterial Pressure (MAP) of more than 25% from baseline
Rates of adverse events and side effects when using TCI for Procedural Sedation in Dentistry - heart rate | Baseline and 5 minute
  A change in the heart rate of more than 25% from baseline
Patient Satisfaction with TCI sedation | Questionnaire presented at baseline ( prior to discharge) and 24 to 48 hours post sedation
  Use of a patient recall and satisfaction questionnaire as a non-technical outcome measure provides researcher/stakeholders with important information on patient's experiences and perspectives
Patient recovery time | Up to 30 minutes
  Measure of time to discharge as defined by the time from last drug administered until patient meets discharge criteria

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Lobb, DDS, Principal Investigator — University of Alberta
Locations (2):
- Dr. Douglas Lobb, Edmonton, Alberta, Canada
- Dr. Don Macalister, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of the study and publication, resulting data, study protocol and other information will be shared.
Supporting Information: CSR
Time Frame: Upon completion of study and publication
Access Criteria: Study protocol, and clinical report